CLINICAL TRIAL: NCT02129231
Title: Ezetimibe/Simvastatin and Rosuvastatin for Oxidative Stress and Mitochondrial Function in Diabetic Polyneuropathy: a Randomized, Double Blinded, Placebo Controlled Clinical Trial
Brief Title: Statins for Oxidative Stress and Mitochondrial Function in Diabetic Polyneuropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Alejandra Guillermina Miranda Diaz, PhD, MD, FACS, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STAT/DPN_2014
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Oxidative Stress; Diabetic Polyneuropathy
Keywords: ezetimibe/simvastatin; rosuvastatin; diabetic polyneuropathy; oxidative stress; mitochondrial dysfunction
MeSH Terms: conditions — Diabetic Neuropathies; Mitochondrial Diseases | interventions — Ezetimibe, Simvastatin Drug Combination; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- placebo (Placebo Comparator): calcined magnesia 100 mg tablets once a day for 16 weeks
  Interventions: Drug: calcined magnesia
- ezetimibe/simvastatin (Active Comparator): ezetimibe/simvastatin 10/20 mg tablets once a day for 16 weeks
  Interventions: Drug: Ezetimibe/simvastatin
- rosuvastatin (Active Comparator): rosuvastatin 20 mg tablets once a day for 16 weeks
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: calcined magnesia — We ensured the patient took the drug at night before meals
  Other Names: placebo
  Arms: placebo
Drug: Ezetimibe/simvastatin — We ensured the patient took the drug at night before meals
  Other Names: Zintrepid; Vytorin
  Arms: ezetimibe/simvastatin
Drug: Rosuvastatin — We ensured the patient took the drug at night before meals
  Other Names: Crestor
  Arms: rosuvastatin

SUMMARY:
Aims: To evaluate the effect of ezetimibe/simvastatin and rosuvastatin on oxidative stress and mitochondrial function in patients with DPN.

Methods: We performed a randomized, double-blinded, placebo-controlled phase II clinical trial in adult patients with type 2 Diabetes Mellitus (T2DM) who had Diabetic Polyneuropathy (DPN) evaluated by composite scores and nerve conduction studies (NCS), HBA1C <12% (108 mmol/mol), previous exclusion of other neuropathies. Ninety-eight persons with T2DM were allocated 1:1:1 to either placebo, ezetimibe/simvastatin 10/20 mg or rosuvastatin 20 mg for 16 weeks, and healthy controls (not randomized) were included for comparisons. Primary outcomes were lipid peroxidation (LPO), nitric oxide (NO), and total antioxidant capacity (TAC); secondary were clinical, NCS and metabolic parameters. Results were expressed as mean ± standard deviation (SD) or standard error of the mean (SEM), frequencies and percentages. Non-parametric analysis was used.

DETAILED DESCRIPTION:
Introduction Nerve dysfunction system in patients with diabetes is known as diabetic neuropathy and is considered as the most prevalent microvascular complication -up to 60%- in type 2 Diabetes Mellitus (T2DM) subjects. Diabetic polyneuropathy (DPN) comprise ≈70% of all cases. Its diagnosis is established by means of validated scores based on clinical features and abnormal nerve conduction studies (NCS). Pathophysiologic findings include loss of multifocal and focal nerve fibers secondary to axonal degeneration an segmental demyelinization, basically due to oxidative stress induced by chronic hyperglycemia, which leads to neural apoptosis. Other mechanisms involved in peripheral nerve injure is nitrosative stress induced by nitric oxide (NO).

Ezetimibe diminishes cholesterol esters content in chylomicrons by reducing liver cholesterol intake which in consequence increases LDL uptake and plasma depuration; as monotherapy it reduces LDL-C by 17%. When combined with simvastatin, cholesterol reduction is potentially increased; furthermore, pleiotropic effects of statins include an increase on nuclear factor kappa B activity and amelioration of superoxide ions after 12 week treatment. Another hydroxy-methyl-glutaryl coenzyme A inhibitor, rosuvastatin, has an antioxidant effect by acting as free radical carrier diminishing mitochondrial and cellular lipid peroxidation (LPO) production.

We conducted this study to evaluate the effect of ezetimibe/simvastatin and rosuvastatin on oxidative stress in patients with DPN.

Methods Study design A randomized, double blinded, placebo controlled phase II clinical trial was performed in the Clinic and Experimental Therapeutics Institute, University of Guadalajara, Mexico. Subjects were assigned to three group treatments in blocks with a parallel sequence 1:1:1 through a randomized computer-based list, generated by a different researcher unaware of drugs given. Patients were divided to: control group that received placebo, ezetimibe/simvastatin and rosuvastatin as a daily single dose for 16 weeks. The selection period was performed from February 2012 to January 2013. We selected 5 non-randomized healthy subjects (HS) from a blood bank to compare the oxidative stress status.

Study population Inclusion criteria were ≥18 years old, T2DM according to American Diabetes Association and DPN by Dyck et. al.3 criteria, HbA1c <12%, and informed consent signed. They were excluded if renal or hepatic failure, pregnant or breastfeeding, other neuropathies (alcohol-induced, radiculopathy, autoimmune, cancer-related), and eliminated if lack treatment adherence (<80% of drug intake), severe adverse drug reaction and/or serious health illness. Patients were selected by invitation in forums; outpatients recruited from primary care clinics; and database collected previously by our Institute from February 2010 to 2012. Patients were instructed to take their drugs only by night at the same time every day, as follows: placebo 100 mg, ezetimibe/simvastatin 10/20 mg, and rosuvastatin 20 mg. All drugs were similar in physical characteristics and presented in dark vials, carefully filled by another group researcher, who placed a respective tag with the patient code. Also, patients were provided with a diary where they would write down the date and time of drug administration, and drug adverse reactions felt. Such information was collected and registered every 4 weeks. Primary outcomes were oxidative stress markers LPO, NO, and TAC before and after 16 week intervention. Secondary outcomes were clinical, NCS and metabolic [fasting glucose, HbA1c, total cholesterol, high and low density lipoproteins (HDL, LDL), and triglycerides] parameters. Safety profile was assessed with drug adverse reactions, renal (urea, creatinin), and hepatic [(alamin- and aspartate-aminotransferase, gama-glutamyltransferase, bilirubins and phosphokinase] laboratory variables.

Oxidative stress and mitochondrial function markers LPO was measured according to kit specifications (Oxford Biomedical Research Inc., FR12), 200 μL of serum where processed with a chromogen substance that reacts with malondialdehyde (MDA) and 4-hydroxy-alkenals (HNA), the absorbance measured at 586 nm, and results expressed in nmol/mL.

Previous deproteinization of the samples, we performed a colorimetric for determining the concentration of NO with 85 µL of serum (Nitric Oxide Assay Kit, User protocol 482650), with results expressed as pmol/mL.

Total antioxidant capacity (TAC) was realized with 200 µL of serum, to obtain values of millimole (mM) equivalent of uric acid (Total Antioxidant Power Kit, No. 02090130, Oxford Biomedical Research®).

Clinical and nerve conduction variables Neuropathic symptoms (NSS) and disability scores (NIS) described by Dyck, et. al. were obtained by physical examination and anamnesis. We also measured the latency, duration, amplitude and motor nerve conduction velocity from fibula, tibial, median and ulnae nerves, and sensitivity parameters from sural, median and ulnae nerves, as required by the American Association of Electrodiagnostic Medicine.

Ethical considerations The study was approved by the Research and Ethics Committee of the Health Science University Center, University of Guadalajara, Mexico. Identification codes were assigned to each participant to guarantee patient confidentiality, and an informed consent form was signed before entering the protocol, according to national and international laws, and also as stipulated by the Helsinki Statements (http://www.wma.net/es/30 publications/ 10 policies/b3/17c.pdf, accessed January 2011).

Statistical analysis The sample size was obtained by a clinical study design formula taking in account a difference change of 0.05 nmol/mL in LPO, 95% confidence interval, 80% potency, and two-tailed p<0.05, which resulted in 21 for each group. Quantitative variables were expressed as mean ± standard deviation. Kolmogorov-Smirnov and Shapiro-Wilk tests were performed to determine the non-parametric distribution of variables. Friedman and Wilcoxon tests were realized for before and after measurements, and Kruskal-Wallis with Mann-Whitney´s U as post-hoc analysis for between group comparisons. Qualitative variables were expressed as frequencies and percentages. Chi square test was used to evaluate differences in dichotomy variables before and after treatment, between group comparisons were determined by Fisher´s exact test and χ2 as needed. Significance level was established with p value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and older
* Type 2 Diabetes Mellitus according to American Diabetes Association
* Diabetic Polyneuropathy by Dyck et. al. criteria
* HbA1c <12%
* Informed consent signed

Exclusion Criteria:

* Renal or hepatic failure
* Pregnant or breastfeeding
* Other neuropathies (alcohol-induced, radiculopathy, autoimmune, cancer-related)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2012-02; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
lipid peroxidation | 16 weeks
  LPO was measured according to kit specifications (Oxford Biomedical Research Inc., FR12), 200 μL of serum where processed with a chromogen substance that reacts with malondialdehyde (MDA) and 4-hydroxy-alkenals (HNA), the absorbance measured at 586 nm, and results expressed in nmol/mL.
Nitric oxide | 16 weeks
  Previous deproteinization of the samples, we performed a colorimetric for determining the concentration of NO with 85 µL of serum (Nitric Oxide Assay Kit, User protocol 482650), with results expressed as pmol/mL.
Total antioxidant capacity | 16 weeks
  Total antioxidant capacity (TAC) was realized with 200 µL of serum, to obtain values of mM equivalent of uric acid (Total Antioxidant Power Kit, No. 02090130, Oxford Biomedical Research®).

SECONDARY OUTCOMES:
neuropathic symptoms score | 16 weeks
  Symptoms referred by the patient as pain and discomfort
neuropathic impairment score | 16 weeks
  Neuropathic signs assessed by the physician through neurological techniques previously published by Dyck et. al.
nerve conduction studies | 16 weeks
  Latency, duration, amplitude and motor nerve conduction velocity from fibula, tibial, median and ulnae nerves, and sensitivity parameters from sural, median and ulnae nerves, as required by the American Association of Electrodiagnostic Medicine.

OTHER OUTCOMES:
Creatinin | 16 weeks
  We measured creatinin to evaluate renal function.
aspartate aminotransferase | 16 weeks
  We measured aspartate aminotransferase regarding hepatic function.
alanine aminotransferase | 16 weeks
  We measured alanine aminotransferase regarding hepatic function.

CONTACTS AND LOCATIONS:
Overall Officials: Luis M Roman-Pintos, PhD, MD, Study Chair — University of Guadalajara; Alejandra G Miranda-Diaz, PhD,MD,FACS, Study Director — University of Guadalajara; Adolfo D Rodriguez-Carrizalez, PhD, MD, Study Chair — University of Guadalajara; Geannyne Villegas-Rivera, PhD, MD, Study Chair — University of Guadalajara
Locations (1):
- Cardiovascular Research Unit, Guadalajara, Jalisco, Mexico

REFERENCES:
- [Background] Hernandez-Ojeda J, Cardona-Munoz EG, Roman-Pintos LM, Troyo-Sanroman R, Ortiz-Lazareno PC, Cardenas-Meza MA, Pascoe-Gonzalez S, Miranda-Diaz AG. The effect of ubiquinone in diabetic polyneuropathy: a randomized double-blind placebo-controlled study. J Diabetes Complications. 2012 Jul-Aug;26(4):352-8. doi: 10.1016/j.jdiacomp.2012.04.004. Epub 2012 May 16. PMID 22595020
- [Derived] Villegas-Rivera G, Roman-Pintos LM, Cardona-Munoz EG, Arias-Carvajal O, Rodriguez-Carrizalez AD, Troyo-Sanroman R, Pacheco-Moises FP, Moreno-Ulloa A, Miranda-Diaz AG. Effects of Ezetimibe/Simvastatin and Rosuvastatin on Oxidative Stress in Diabetic Neuropathy: A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Oxid Med Cell Longev. 2015;2015:756294. doi: 10.1155/2015/756294. Epub 2015 Jul 28. PMID 26290682